CLINICAL TRIAL: NCT06033976
Title: Endoscopic Submucosal Dissection Patients Registry in "Agrippa Ionescu" Hospital, Bucharest, Romania
Brief Title: Endoscopic Submucosal Dissection Registry
Acronym: ESDREG
Status: Recruiting | Type: Observational
Sponsor: Carol Davila University of Medicine and Pharmacy (Other)
Responsible Party: Principal Investigator, Mihai Ciocirlan, Clinical Professor (Associate Professor), Carol Davila University of Medicine and Pharmacy
Other Study IDs: ESDREG
Record Dates: First submitted 2023-09-03; First posted 2023-09-13 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Neoplasm, Stomach; Neoplasm, Colorectal; Neoplasm, Esophagus; Neoplasm, Duodenal
MeSH Terms: conditions — Stomach Neoplasms; Colorectal Neoplasms; Esophageal Neoplasms; Duodenal Neoplasms | interventions — Endoscopic Mucosal Resection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples Without DNA — Resected specimens of the gastrointestinal tract, fixed in formalin
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Endoscopic submucosal dissection (ESD) — Endoscopic injection of fluid into the gastrointestinal submucosal space followed by endoscopic knife dissection around and under the lesion so as to remove the lesion specimen in one piece with lesion free resection margins.
  Other Names: ESD

SUMMARY:
This is a patient registry for all cases of pre-neoplastic or early neoplastic digestive tract lesions treated with curative intention by endoscopic submucosal dissection (ESD) technique.

DETAILED DESCRIPTION:
Cases will be registered one by one in an electronic record, with the consent of the patient and respecting all legal requirements.

ELIGIBILITY:
Inclusion Criteria:

* epithelial pre-neoplastic (eg. adenoma, dysplasia) lesion on the esophageal, gastric, duodenal or colorectal mucosa
* non-epithelial (eg. neuroendocrine tumor) lesion on the esophageal, gastric, duodenal or colorectal mucosa
* age > 18 years old
* informed consent

Exclusion Criteria:

* age < 18 years old
* no informed consent

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed at or referred to Gastroenterology Clinic, University of Medicine and Pharmacy, "Agrippa Ionescu" Hospital, Bucharest, Romania
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2031-01 (Estimated); Study Completion 2031-01 (Estimated)

PRIMARY OUTCOMES:
Rate of curative resection | through study completion, an average of 1 year

SECONDARY OUTCOMES:
Rate of R0 resection | through study completion, an average of 1 year

OTHER OUTCOMES:
Rate of perforation | 30 days
Rate of delayed bleeding | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Mihai L Ciocirlan, Associate Professor, Principal Investigator — Carol Davila University of Medicine and Pharmacy
Locations (1):
- "Agrippa Ionescu" Hospital, Bucharest, Romania

IPD SHARING:
Plan to Share IPD: No